CLINICAL TRIAL: NCT03141346
Title: Home Intervention for Reducing Sugary Drinks and Obesity in Hispanic Women-infants
Brief Title: Improving the Eating Habits of Mother and Her Infant Via Sugar Reduction
Acronym: MAMITA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Michael I. Goran, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHLA-18-00571
Record Dates: First submitted 2017-05-01; First posted 2017-05-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Obesity
Keywords: mother; infant; nutrition; sugar; obesity; growth
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): A control health education program to promote general health and safety
  Interventions: Behavioral: Control health education program
- Sugar Reduction Program Only (Experimental): A health education program that focuses on sugar reduction
  Interventions: Behavioral: Sugar reduction health education program
- Sugar Reduction Program & Water Delivery (Experimental): A health education program that focuses on sugar reduction and provides home bottled water delivery
  Interventions: Behavioral: Sugar reduction health education program; Other: Home water delivery

INTERVENTIONS:
Behavioral: Sugar reduction health education program — A health education program incorporating sugar reduction education and monitoring provided by a trained health educator over 24 months. The intervention program will be delivered by the health educator during in-person home visits, or virtually via phone or video calls.
  Arms: Sugar Reduction Program & Water Delivery; Sugar Reduction Program Only
Behavioral: Control health education program — Control health education program provided by a trained health educator over 24 months. The intervention program will be delivered by the health educator during in-person home visits, or virtually via phone or video calls.
  Arms: Control
Other: Home water delivery — Home delivery of bottled water administered over 24 months
  Arms: Sugar Reduction Program & Water Delivery

SUMMARY:
The purpose of this study is to determine whether a health education program incorporating sugar sweetened beverage and juice (SSB/J) reduction and home water delivery affects maternal and infant risk for obesity by randomizing mother-infant dyads to one of three 24-month interventions: Group 1 (control): standard health education program only; Group 2 (translation): health education program focused on sugar reduction; and Group 3 (efficacy): health education program focused on sugar reduction and bottled water delivery. The intervention program will be delivered by trained health educators during in-person home visits, or virtually via phone or video calls.

DETAILED DESCRIPTION:
This study will determine whether a health education program incorporating sugar sweetened beverage and juice (SSB/J) reduction and home water delivery affects maternal and infant risk for obesity. The postpartum period is a time of both opportunity and vulnerability for mothers and their infants to diminish risk for obesity and related health problems. This is particularly relevant in the context of Hispanic families. Hispanic mothers are at high-risk for excess gestational weight gain and postpartum weight retention, and their infants are at high-risk for rapid weight gain associated with early onset obesity. A contributing factor may be their intake of SSB/J. There is a high prevalence of reported SSB/J consumption in low-income Hispanic households, and Hispanic mothers are more likely to incorporate sweet foods during weaning. Because evidence suggests that obese Hispanic children are responsive to SSB/J reduction and substitution with non-caloric beverages, this may be a potential strategy for Hispanic mothers that may also be beneficial for their infants.

This study will be conducted in Los Angeles. Two-hundred-and-forty Hispanic mothers and their infants will be recruited. They will be randomly assigned to: group 1, a standard health education program only; group 2, a health education program that incorporates sugar reduction; and group 3, a health education program that incorporates sugar reduction with home bottled water delivery. The intervention program will be delivered by trained health educators during in-person home visits, or virtually via phone or video calls. The main outcomes are maternal weight status and infant weight change. We will also assess maternal and infant diet using 24-hour recalls, and maternal feeding style and infant eating behaviors using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who self-identify as Hispanic
* Mothers who have or have had singleton births
* Mothers will be recruited prior to their infant's birth or up to 1-month postpartum
* Mothers must be able/willing to understand the procedures of the study, and must be able to read English or Spanish at a 5th grade level
* Mothers who are habitual consumers of sugar sweetened beverages and juices

Exclusion Criteria:

* Physician diagnosis of a major medical illness (including type 1 or type 2 diabetes) or eating disorder in mothers
* Physical, mental, or cognitive issues that prevent participation
* Chronic use of any medication that may affect body weight or composition, insulin resistance, or lipid profiles
* Current smoking (more than 1 cigarette in the past week) or use of other recreational drugs
* Clinical diagnosis of gestational diabetes
* Pre-term/low birth weight infants, or diagnosis of any fetal abnormalities
* Mothers less than 18 years of age at the time of delivery will not be eligible as to avoid potential confounding from those subjects who might still be completing adolescent growth

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 211 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Maternal height at baseline | Baseline
  Height (cm) will be measured using a stadiometer.
Maternal height at 6 months | 6 months
  Height (cm) will be measured using a stadiometer.
Maternal height at 12 months | 12 months
  Height (cm) will be measured using a stadiometer.
Maternal height at 24 months | 24 months
  Height (cm) will be measured using a stadiometer.
Maternal weight at baseline | Baseline
  Weight (kg) will be measured using a portable digital scale.
Maternal weight at 6 months | 6 months
  Weight (kg) will be measured using a portable digital scale.
Maternal weight at 12 months | 12 months
  Weight (kg) will be measured using a portable digital scale.
Maternal weight at 24 months | 24 months
  Weight (kg) will be measured using a portable digital scale.
Maternal BMI at baseline | Baseline
  Body Mass Index (BMI) will be calculated based on the equation (weight in kg)/(height in m)^2.
Maternal BMI at 6 months | 6 months
  Body Mass Index (BMI) will be calculated based on the equation (weight in kg)/(height in m)^2.
Maternal BMI at 12 months | 12 months
  Body Mass Index (BMI) will be calculated based on the equation (weight in kg)/(height in m)^2.
Maternal BMI at 24 months | 24 months
  Body Mass Index (BMI) will be calculated based on the equation (weight in kg)/(height in m)^2.
Infant length at baseline | Baseline
  Infant length (cm) will be measured using an infant measure mat.
Infant length at 6 months | 6 months
  Infant length (cm) will be measured using an infant measure mat.
Infant length at 12 months | 12 months
  Infant length (cm) will be measured using an infant measure mat.
Infant length at 24 months | 24 months
  Infant length (cm) will be measured using an infant measure mat.
Infant weight at baseline | Baseline
  Infant weight (kg) will measured using a portable digital scale. For infants that need to be held, weight will be calculated as follows: (combined mother + infant weight) - (mother only weight).
Infant weight at 6 months | 6 months
  Infant weight (kg) will measured using a portable digital scale. For infants that need to be held, weight will be calculated as follows: (combined mother + infant weight) - (mother only weight).
Infant weight at 12 months | 12 months
  Infant weight (kg) will measured using a portable digital scale. For infants that need to be held, weight will be calculated as follows: (combined mother + infant weight) - (mother only weight).
Infant weight at 24 months | 24 months
  Infant weight (kg) will measured using a portable digital scale. For infants that need to be held, weight will be calculated as follows: (combined mother + infant weight) - (mother only weight).
Infant weight z-scores at baseline | Baseline
  Weight and length will be used to calculate weight-for-length (WLZ) and weight-for-age (WAZ) z-scores using the WHO Child Growth Standards, as recommended by the CDC for children <24 mos.
Infant weight z-scores at 6 months | 6 months
  Weight and length will be used to calculate weight-for-length (WLZ) and weight-for-age (WAZ) z-scores using the WHO Child Growth Standards, as recommended by the CDC for children <24 mos.
Infant weight z-scores at 12 months | 12 months
  Weight and length will be used to calculate weight-for-length (WLZ) and weight-for-age (WAZ) z-scores using the WHO Child Growth Standards, as recommended by the CDC for children <24 mos.
Infant weight z-scores at 24 months | 24 months
  Weight and length will be used to calculate weight-for-length (WLZ) and weight-for-age (WAZ) z-scores using the WHO Child Growth Standards, as recommended by the CDC for children <24 mos.
Infant body fat measured using an EchoMRI body composition analyzer at baseline | Baseline
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant body fat in grams.
Infant body fat measured using an EchoMRI body composition analyzer at 6 months | 6 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant body fat in grams.
Infant body fat measured using an EchoMRI body composition analyzer at 12 months | 12 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant body fat in grams.
Infant body fat measured using an EchoMRI body composition analyzer at 24 months | 24 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant body fat in grams.
Infant lean mass measured using an EchoMRI body composition analyzer at baseline | Baseline
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant lean mass in grams.
Infant lean mass measured using an EchoMRI body composition analyzer at 6 months | 6 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant lean mass in grams.
Infant lean mass measured using an EchoMRI body composition analyzer at 12 months | 12 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant lean mass in grams.
Infant lean mass measured using an EchoMRI body composition analyzer at 24 months | 24 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant lean mass in grams.
Infant total body water measured using an EchoMRI body composition analyzer at baseline | Baseline
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant total body water in grams.
Infant total body water measured using an EchoMRI body composition analyzer at 6 months | 6 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant total body water in grams.
Infant total body water measured using an EchoMRI body composition analyzer at 12 months | 12 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant total body water in grams.
Infant total body water measured using an EchoMRI body composition analyzer at 24 months | 24 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant total body water in grams.
Infant free body water measured using an EchoMRI body composition analyzer at baseline | Baseline
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant free body water in grams.
Infant free body water measured using an EchoMRI body composition analyzer at 6 months | 6 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant free body water in grams.
Infant free body water measured using an EchoMRI body composition analyzer at 12 months | 12 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant free body water in grams.
Infant free body water measured using an EchoMRI body composition analyzer at 24 months | 24 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant free body water in grams.

SECONDARY OUTCOMES:
Maternal pregravid BMI | Baseline
  Maternal BMI prior to pregnancy will be derived from pregravid BMI (recall during pregnancy at baseline visit) using the equation (weight in kg)/(height in m)^2.
Maternal blood pressure at baseline | Baseline
  Sitting blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal blood pressure at 6 months | 6 months
  Sitting blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal blood pressure at 12 months | 12 months
  Sitting blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal blood pressure at 24 months | 24 months
  Sitting blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal resting heart rate at baseline | Baseline
  Sitting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal resting heart rate at 6 months | 6 months
  Sitting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal resting heart rate at 12 months | 12 months
  Sitting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal resting heart rate at 24 months | 24 months
  Sitting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal diet at baseline | Baseline
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Maternal diet at 6 months | 6 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Maternal diet at 12 months | 12 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Maternal diet at 24 months | 24 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Infant diet at 6 months | 6 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Mothers will be interviewed to report on their infant's food intake, starting at the 6-month visit when infants are likely to be introduced to solid foods. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Infant diet at 12 months | 12 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Mothers will be interviewed to report on their infant's food intake, starting at the 6-month visit when infants are likely to be introduced to solid foods. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Infant diet at 24 months | 24 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Mothers will be interviewed to report on their infant's food intake, starting at the 6-month visit when infants are likely to be introduced to solid foods. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Infant feeding score assessed by Infant Feeding Questionnaire at baseline | Baseline
  Infant feeding score will be assessed using the Baughcum Infant Feeding Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: concern about the child undereating or becoming underweight; concern about infant's hunger; awareness of infant's cues; concern about the infant becoming overweight or overeating; feeding the infant on schedule; using food to calm the infant; social interaction during feeding.
Infant feeding score assessed by Infant Feeding Questionnaire at 6 months | 6 months
  Infant feeding score will be assessed using the Baughcum Infant Feeding Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: concern about the child undereating or becoming underweight; concern about infant's hunger; awareness of infant's cues; concern about the infant becoming overweight or overeating; feeding the infant on schedule; using food to calm the infant; social interaction during feeding.
Infant feeding score assessed by Infant Feeding Questionnaire at 12 months | 12 months
  Infant feeding score will be assessed using the Baughcum Infant Feeding Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: concern about the child undereating or becoming underweight; concern about infant's hunger; awareness of infant's cues; concern about the infant becoming overweight or overeating; feeding the infant on schedule; using food to calm the infant; social interaction during feeding.
Infant feeding score assessed by Infant Feeding Questionnaire at 24 months | 24 months
  Infant feeding score will be assessed using the Baughcum Infant Feeding Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: concern about the child undereating or becoming underweight; concern about infant's hunger; awareness of infant's cues; concern about the infant becoming overweight or overeating; feeding the infant on schedule; using food to calm the infant; and social interaction during feeding.
Infant feeding style score assessed by Infant Feeding Style Questionnaire at baseline | Baseline
  Infant feeding style score will be assessed using the Thompson Infant Feeding Style Questionnaire. Questions are scored using the following scale: 1-5; disagree, slightly disagree, neutral, slightly agree, agree. Average scores will be used to determine the following constructs: laissez-faire; pressuring; restrictive; responsive; and indulgent.
Infant feeding style score assessed by Infant Feeding Style Questionnaire at 6 months | 6 months
  Infant feeding style score will be assessed using the Thompson Infant Feeding Style Questionnaire. Questions are scored using the following scale: 1-5; disagree, slightly disagree, neutral, slightly agree, agree. Average scores will be used to determine the following constructs: laissez-faire; pressuring; restrictive; responsive; and indulgent.
Infant feeding style score assessed by Infant Feeding Style Questionnaire at 12 months | 12 months
  Infant feeding style score will be assessed using the Thompson Infant Feeding Style Questionnaire. Questions are scored using the following scale: 1-5; disagree, slightly disagree, neutral, slightly agree, agree. Average scores will be used to determine the following constructs: laissez-faire; pressuring; restrictive; responsive; and indulgent.
Infant feeding style score assessed by Infant Feeding Style Questionnaire at 24 months | 24 months
  Infant feeding style score will be assessed using the Thompson Infant Feeding Style Questionnaire. Questions are scored using the following scale: 1-5; disagree, slightly disagree, neutral, slightly agree, agree. Average scores will be used to determine the following constructs: laissez-faire; pressuring; restrictive; responsive; and indulgent.
Infant behavior score assessed by Infant Behavior Questionnaire at baseline | Baseline
  Infant behavior score will be assessed using the Rothbart Infant Behavior Questionnaire. Questions are scored using the following scale: 1-7; never, very rarely, less than half the time, about half the time, more than half the time, almost always, always. Composite scores will be used to determine the following constructs: surgency/extroversion; negative affectivity; and orienting/regulation.
Infant behavior score assessed by Infant Behavior Questionnaire at 6 months | 6 months
  Infant behavior score will be assessed using the Rothbart Infant Behavior Questionnaire. Questions are scored using the following scale: 1-7; never, very rarely, less than half the time, about half the time, more than half the time, almost always, always. Composite scores will be used to determine the following constructs: surgency/extroversion; negative affectivity; and orienting/regulation.
Infant behavior score assessed by Early Child Behavior Questionnaire at 12 months | 12 months
  Infant behavior score will be assessed using the Rothbart Early Child Behavior Questionnaire. Questions are scored using the following scale: 1-7; never, very rarely, less than half the time, about half the time, more than half the time, almost always, always. Composite scores will be used to determine the following constructs: negative affectivity; surgency-extroversion; and effortful control.
Infant behavior score assessed by Early Child Behavior Questionnaire at 24 months | 24 months
  Infant behavior score will be assessed using the Rothbart Early Child Behavior Questionnaire. Questions are scored using the following scale: 1-7; never, very rarely, less than half the time, about half the time, more than half the time, almost always, always. Composite scores will be used to determine the following constructs: negative affectivity; surgency-extroversion; and effortful control.
Infant eating behavior score assessed by Baby Eating Behavior Questionnaire at baseline | Baseline
  Infant eating behavior score will be assessed using the Llewellyn Baby Eating Behavior Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: food responsiveness; satiety responsiveness; slowness in eating; enjoyment of food; and general appetite.
Infant eating behavior score assessed by Baby Eating Behavior Questionnaire at 6 months | 6 months
  Infant eating behavior score will be assessed using the Llewellyn Baby Eating Behavior Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: food responsiveness; satiety responsiveness; slowness in eating; enjoyment of food; and general appetite.
Infant eating behavior score assessed by Child Eating Behavior Questionnaire at 12 months | 12 months
  Infant eating behavior score will be assessed using the Wardle Child Eating Behavior Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: food responsiveness; enjoyment of food; emotional overeating; desire to drink; satiety responsiveness; slowness in eating; emotional undereating; and fussiness.
Infant eating behavior score assessed by Child Eating Behavior Questionnaire at 24 months | 24 months
  Infant eating behavior score will be assessed using the Wardle Child Eating Behavior Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: food responsiveness; enjoyment of food; emotional overeating; desire to drink; satiety responsiveness; slowness in eating; emotional undereating; and fussiness.
Breast milk composition at baseline | Baseline
  Breast milk will be collected from mothers at least 1½ hours since the last feeding and while the mother has fasted at least 1 hour. Samples will be analyzed for glucose, fructose, galactose, lactose and sucrose by mass spectrometry. Samples will be available for analysis of insulin, leptin, and energy content.
Breast milk composition at 6 months | 6 months
  Breast milk will be collected from mothers at least 1½ hours since the last feeding and while the mother has fasted at least 1 hour. Samples will be analyzed for glucose, fructose, galactose, lactose and sucrose by mass spectrometry. Samples will be available for analysis of insulin, leptin, and energy content.
Breast milk composition at 12 months | 12 months
  Breast milk will be collected from mothers at least 1½ hours since the last feeding and while the mother has fasted at least 1 hour. Samples will be analyzed for glucose, fructose, galactose, lactose and sucrose by mass spectrometry. Samples will be available for analysis of insulin, leptin, and energy content.
Breast milk composition at 24 months | 24 months
  Breast milk will be collected from mothers at least 1½ hours since the last feeding and while the mother has fasted at least 1 hour. Samples will be analyzed for glucose, fructose, galactose, lactose and sucrose by mass spectrometry. Samples will be available for analysis of insulin, leptin, and energy content.

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Goran, Principal Investigator — University of Southern California; Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Machle CJ, Berger PK, Salvy SJ, Rios C, Durazo-Arvizu R, Goran MI. Efficacy of a 24-month behavioral intervention focused on sugary beverage reduction for Latino mother-infant dyads: evidence from a randomized controlled trial. Am J Clin Nutr. 2025 Feb;121(2):355-366. doi: 10.1016/j.ajcnut.2024.11.009. Epub 2025 Jan 9. PMID 39909707